CLINICAL TRIAL: NCT03529890
Title: A Prospective, Single Arm, Multicenter, Phase II-Trial to Assess Safety and Efficacy of Preoperative RAdiation Therapy Before Radical CystEctomy Combined With ImmunoTherapy in Locally Advanced Urothelial Carcinoma of the Bladder
Brief Title: Radio-Immunotherapy Before Cystectomy in Locally Advanced Urothelial Carcinoma of the Bladder
Acronym: RACE IT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Technical University of Munich (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB 65/18; CA209-9WT (Other Grant/Funding Number: BMS)
Record Dates: First submitted 2018-03-26; First posted 2018-05-18 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2021-12

CONDITIONS: Urinary Bladder Cancer
Keywords: locally advanced urothelial carcinoma; immunotherapy; cystectomy; radiation; nivolumab
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Nivolumab; Cystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radio-Immunotherapy before cystectomy (Experimental): Single arm treatment with Nivolumab during a neoadjuvant radiation therapy of the pelvis before radical cystectomy with standardized pelvic lymphadenectomy
  Interventions: Drug: Nivolumab; Radiation: Radiation therapy of the pelvis; Procedure: Radical cystectomy with standardized pelvic lymphadenectomy

INTERVENTIONS:
Drug: Nivolumab — Experimental intervention:
  Immunotherapy with 4 cycles of Nivolumab: 240 mg intravenously every 2 weeks, starting one week before radiotherapy (week1, d1), last infusion on week 7, d1
  Other Names: Opdivo
Radiation: Radiation therapy of the pelvis — Neoadjuvant radiation therapy of pelvis with 45+5,4 Gy for 6 weeks: 28 x 1.8 Gy including a boost of bladder with 5.4 Gy, starting with week 2 (d1)
Procedure: Radical cystectomy with standardized pelvic lymphadenectomy — Radical cystectomy with standardized bilateral pelvic lymphadenectomy: performed between week 11 - 15 (Aim: week 13)

SUMMARY:
A prospective, single arm, multicenter, Phase II-Trial to assess safety and efficacy of preoperative Radiation therapy before radical CystEctomy combined with ImmunoTherapy in locally advanced urothelial carcinoma of the bladder

DETAILED DESCRIPTION:
Patients with locally advanced bladder cancer have a poor prognosis despite radical surgical therapy. The addition of perioperative combination chemotherapy did not add significant benefit to surgery alone. There is data indicating a synergistic effect of radiation and immunotherapy. Therefore, combined application of radiotherapy with Nivolumab before radical cystectomy might lead to improved cure rates and local control in this poor prognosis group with locally advanced bladder cancer. The aim of this phase-II study is to assess feasibility and safety of immunotherapy combined with neoadjuvant radiation before radical cystectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, locally advanced bladder cancer (cT3/4 cN0/N+ cM0)

   1. Urothelial cancer with at least 10% urothelial differentiation (excluding presence of small cell differentiation, which is not allowed in any percentage)
   2. Histologic proof of muscle invasion in TUR-B specimen: ≥ pT2
   3. Signs of locally advanced bladder cancer (at least one of the following must apply):

   i. cT3/4 in imaging studies (bladder wall thickening or infiltration of perivesical fat/adjacent organs)

   ii. Presence of hydronephrosis (or status post nephrostomy/ureteral stent due to hydronephrosis)

   iii. Pelvic lymph nodes ≥ 8 mm in short axis
2. Ineligibility for neoadjuvant cisplatin-based chemotherapy due to any of the following criteria:

   1. Creatinine Clearance (using the Cockcroft-Gault formula) < 60 mL/min
   2. Hearing loss ≥ grade 2 (CTCAE version 4)
   3. Peripheral neuropathy ≥ grade 2 (CTCAE version 4)
   4. ECOG performance score 2
3. Subjects that are eligible for cisplatin may be candidates if they refuse available neoadjuvant cisplatin-based chemotherapy, despite being informed by the investigator about the treatment options. The subject's refusal must be thoroughly documented.
4. Eligible for radical cystectomy
5. ECOG 0 - 2
6. Estimated life expectancy > 6 months
7. Adequate function of bone marrow, liver and kidney:

   1. WBC ≥ 2000/μL
   2. Neutrophils ≥ 1500/μL
   3. Platelets ≥ 100 × 103/μL
   4. Hemoglobin ≥ 9.0 g/dL
   5. AST ≤ 3 × ULN
   6. ALT ≤ 3 × ULN
   7. Total bilirubin ≤ 1.5 × ULN (except in participants with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
   8. GFR ≥ 15 mL/min without hydronephrosis. In case of hydronephrosis, drainage should be performed prior to inclusion preferably by nephrostomy, alternatively by ureteral stent placement. Use measured creatinine-clearance or estimated clearance (Cockcroft-Gault formula):
   9. Female CrCl = [(140 - age in years) × weight in kg × 0.85] / [72 x serum creatinine in mg/dL] ii. Male CrCl = [(140 - age in years) × weight in kg × 1.00] / [72 x serum creatinine in mg/dL]
8. Informed consent:

   1. Participants must have signed and dated an IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal participant care.
   2. Participants must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, and other requirements of the study
9. Body weight 35 kg - 160 kg
10. Female patients with childbearing potential must have a negative serum pregnancy test prior to start of trial.
11. Women of childbearing potential (WOCBP) and men (who are sexually active with WOCBP) must use any contraceptive method with a failure rate of less than 1% per year (see Appendix 15.7). These patients will be instructed to adhere to contraception for the period between inclusion into the study and surgery (which leads to sterility). Women who are not of childbearing potential (i.e. who are postmenopausal or surgically sterile) as well as sterile men do not require contraception. If patients do not undergo surgery or in the rare case of fertility preserving cystectomy , effective contraception should be used for at least 5 months following the last dose of Nivolumab. In the latter instance serum pregnancy testing is required in WOCBP at the end of the 5 months.

Exclusion Criteria:

1. Metastatic disease defined as distant metastasis or suspicious lymph nodes (> 10mm short axis) outside the pelvis (clearly above aortic bifurcation) using RECIST 1.1 criteria. Enlarged lymph nodes in the pelvis below or at aortic bifurcation are NO exclusion criterion irrespective of size.
2. Prior chemotherapy before treatment (not including intravesical chemotherapy)
3. Prior radiation therapy of the pelvis
4. Active, known or suspected autoimmune disease (not including: vitiligo, allergic rhinitis/asthma, type 1 diabetes mellitus, residual hypothyroidism due to an autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger)
5. Immunosuppressive treatment with corticosteroids or other drugs within 14 days of study drug administration (not including: inhaled or topical steroids and adrenal replacement doses are permitted in the absence of active autoimmune disease)
6. Experimental therapy or clinical trial at time of inclusion or the previous 4 weeks
7. Previous treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways (not including BCG therapy)
8. Any uncontrolled or severe cardiovascular or pulmonary disease determined by the investigator, including i) NYHA functional classification III or IV, congestive heart failure, unstable or poorly controlled angina, uncontrolled hypertension, serious arrhythmia or myocardial infarction in previous 12 months before inclusion; ii) Subjects with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxic.
9. End-stage kidney disease defined as GFR < 15ml/min or need for dialysis in absence of hydronephrosis. In case of hydronephrosis, drainage should be performed prior to inclusion preferably by nephrostomy, alternatively by ureteral stent placement.
10. Thromboembolic events like pulmonary embolism or apoplexy in previous 3 months
11. Other active tumor disease (not including basal cell carcinoma of the skin, carcinoma in situ of the cervix and incidental prostate carcinoma). Tumor is regarded non active after curative therapy and 5 years of follow up without pathological findings.
12. Medium to extended surgery or trauma in the previous 4 weeks (not including transurethral bladder resection, nephrostomy or ureteral stent or biopsy)
13. Uncontrolled and serious somatic or mental illness
14. Age < 18 years
15. Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.
16. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities [§ 40 Abs. 1 S. 3 Nr. 4 AMG].
17. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG].
18. Female subjects who are pregnant, breast-feeding or male/female patients of childbearing potential who are not employing an effective method of birth control (failure rate of less than 1% per year). [Acceptable methods of contraception are: implants, injectable contraceptives, combined oral contraceptives, intrauterine pessaries (only hormonal devices), sexual abstinence or vasectomy of the partner, see Appendix 15.7.].
19. Participation in another clinical study with an investigational product during the last 30 days before inclusion or 7 half-lifes of previously used trial medication, whichever is longer.
20. Hypersensitivity to Nivolumab or any of it's excipients.
21. Prior organ transplantation
22. Positive test result for hepatitis B or C indicating acute or chronic infection.
23. Positiv HIV test or acquired immunodeficiency syndrome (AIDS)
24. Serious or uncontrolled medical disorder or active infection that, in the opinion of the investigator, may increase the risk associated with study participation, study drug administration, or would impair the ability of the patient to receive protocol therapy
25. Gastrointestinal disorders, particularly those with high risk of perforation or fistula formation including i) active peptic ulcer disease or active inflammatory bowel disease (incl. ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis during screening and/or ii) history of abdominal fistula or bowel perforation within 6 months prior to first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2019-02-04 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with completed Treatment | end of week 15
  Completed Treatment (consisting of radio-immunotherapy and radical cystectomy) is defined by Administration of at least 2 complete cycles of nivolumab 240 mg and Administration of at least 23 of planned 28 Radiation fractions (at least 41.4 Gy in total)

SECONDARY OUTCOMES:
Acute toxicity of preoperative radio-immunotherapy | beginning of treatment until 3 months after end of therapy
  according to CTCAE v4, typical predefined side effects of surgery will be excluded from analysis
Rate of immune related toxicities | beginning of treatment until 12 months after cystectomy
  immune mediated pneumonitis, colitis, Hepatitis, hypophysitis, adrenal insufficiency, hypo-/hyperthyroidism, Diabetes (type 1), Nephritis, Skin reactions
Late toxicity | 3 months after end of therapy until 12 months after cystectomy
  according to CTCAE v4
Disease free survival | until 12 months after cystectomy
  defined by local recurrence or distant metastasis dor death in R0 resected patients during 1 year follow
Overall survival | until 12 months after cystectomy
  time to death by any cause
radiological Overall Response rate | after completion of radioimmunotherapy before cystectomy (week 12; range 11-14)
  complete Remission, partial Remission, stable disease, progressive disease
ypT0 rate | after cystectomy was performed (week 16)
  rate of pT0 after therapy
surgical margin Status | after cystectomy was performed (week 16)
  R0, R1, R2

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian C Schmid, PD Dr. med, Principal Investigator — Department of Urology, Klinikum rechts der Isar der Technischen Universität München
Locations (3):
- Germany (3):
  - Department of Urology, Klinikum rechts der Isar der Technischen Universität München, München
  - Universitätsklinikum Ulm; Klinik für Urologie, Ulm
  - Department of Urology, Universitätsklinikum Würzburg, Würzburg

REFERENCES:
- [Derived] Schmid SC, Koll FJ, Rodel C, Maisch P, Sauter A, Beckert F, Seitz A, Kubler H, Flentje M, Chun F, Combs SE, Schiller K, Gschwend JE, Retz M. Radiation therapy before radical cystectomy combined with immunotherapy in locally advanced bladder cancer - study protocol of a prospective, single arm, multicenter phase II trial (RACE IT). BMC Cancer. 2020 Jan 3;20(1):8. doi: 10.1186/s12885-019-6503-6. PMID 31900121